CLINICAL TRIAL: NCT04495595
Title: Influence of the Biological Maturation on the Antrhopometric Variables and Sport Performance in Volleyball Players
Status: Completed | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Mario Albaladejo-Saura, Principal Investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: CE061921
Record Dates: First submitted 2020-07-23; First posted 2020-08-03 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Development, Adolescent; Body Weight Changes
Keywords: Sport performance; Volleyball; Anthropometry; Biological maturation
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There is no intervention due to the observational, cross-sectional design of the study

SUMMARY:
The project consists of a cross-sectional study in which anthropometric variables, general and specific performance variables of volleyball will be measured, and the biological maturity stage will be calculated. The main objective is to establish a relationship between the biological maturation state, the anthropometric characteristics and the performance in physical fitness tests in volleyball players between 12 and 15 years of age. To do this, there will be all the clubs in the Region of Murcia that have federated teams in these categories.

ELIGIBILITY:
Inclusion Criteria:

* To play volleyball in a regular basis
* To have between 12 and 15 years
* To participate in volleiball competitions with the team

Exclusion Criteria:

* To be injured in the moment of the measurement session
* To have skipped most of the training sessions the last month
* To have less than a year of experience playing volleyball

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The sample objetive of the present study are all the volleyball players of Región of Murcia, Spain, that meet the inclusion criteria and voluntarily decide to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Volleyball performance | through study completion, an average of 1 year
  Qualitative assessement of the individual sport performance, taking on account the team position on the league and the role of the player in the team. The instrument used to assess this variable will be a questionnaire and the result will be expressed in points (1 to 5 points).
Biological maturation | through study completion, an average of 1 year
  Calculated with anthropometric variables. The result obtained indicates the time left to the growth peak or the time that has passed from the growth peak
Muscle mass | through study completion, an average of 1 year
  Muscle mass will be assessed with the corresponding formulas. The result will be expressed in kilograms
Fat mass | through study completion, an average of 1 year
  Fat mass will be assessed with the corresponding formulas. The result will be expressed in kilograms
Bone mass | through study completion, an average of 1 year
  Bone mass will be assessed with the corresponding formulas. The result will be expressed in kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No